CLINICAL TRIAL: NCT03263299
Title: Value of Cabergoline and Low Dose Aspirin in Poor Responders Undergoing ICSI-ET Using Microdose GnRH Agonist Flare-Up-Protocol
Brief Title: Value of Cabergoline and Low Dose Aspirin in Poor Responders Undergoing ICSI-ET With GnRH Agonist Flare-Up-Protocol
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Invitro Fertilization
MeSH Terms: interventions — Cabergoline; Aspirin; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- cabergoline group (Active Comparator): received cabergoline in addition to aspirin. Cabergoline was administered in a dose of 1 mg/week in two divided doses which was terminated after embryo transfer. Aspirin was administered in daily dose of 80 mg initiated at the start of down-regulation with luteal leuprolide
  Interventions: Drug: cabergoline; Drug: Aspirin; Drug: GnRH agonist
- Aspirin group (Active Comparator): Aspirin was administered in daily dose of 80 mg initiated at the start of down-regulation with luteal leuprolide
  Interventions: Drug: Aspirin; Drug: GnRH agonist
- GnRH Group (Active Comparator): Microdose flare-up regimen. The patient received diluted doses of the GnRH agonist leuprolide acetate 40 µg, given subcutaneously twice daily. Two days later, stimulation is initiated by intramuscular (IM) injections of HMG (Merional, IBSA, Germany) in a dose of 300 IU/day.
  Interventions: Drug: GnRH agonist

INTERVENTIONS:
Drug: cabergoline — Cabergoline was administered in a dose of 1 mg/week in two divided doses which was terminated after embryo transfer
  Arms: cabergoline group
Drug: Aspirin — Aspirin was administered in daily dose of 80 mg initiated at the start of down-regulation with luteal leuprolide
  Arms: Aspirin group; cabergoline group
Drug: GnRH agonist — Microdose flare-up regimen. The patient received diluted doses of the GnRH agonist leuprolide acetate 40 µg, given subcutaneously twice daily. Two days later, stimulation is initiated by intramuscular (IM) injections of HMG (Merional, IBSA, Germany) in a dose of 300 IU/day.

SUMMARY:
Ovarian stimulation will be done using the Microdose flare-up regimen. The patient will receive diluted doses of the GnRH agonist leuprolide acetate 40 µg, given subcutaneously twice daily. Two days later, stimulation will be initiated by intramuscular (IM) injections of HMG (Merional, IBSA, Germany) in a dose of 300 IU/day.

Follicular monitoring began from the ninth day of the cycle by serial vaginal ultrasonography and measurement of serum E2 levels. IM injections of 10000 IU HCG (Choriomon; IBSA, Germany) will be injected when at least 2 follicles 18 mm were observed on ultrasonography.

Oocytes willbe retrieved 36 hours after hCG injection using a 17-gauge aspiration needle under transvaginal ultrasound guidance. The pelvis is evaluated with ultrasound to ensure that there is no internal bleeding.

After fertilization was confirmed when two polar bodies and two pronuclear were observed 18-20 hours after insemination, one to three grade A embryos were transferred at day 3 fertilization.

The luteal phase support will be initiated from the day of oocyte retrieval for all patients with (Cyclogest 400 mg, Actavis pharmaceutical, UK) vaginal suppositories per day till the day of serum pregnancy test was done.

DETAILED DESCRIPTION:
Ovarian stimulation was done using the Microdose flare-up regimen. The patient received diluted doses of the GnRH agonist leuprolide acetate 40 µg, given subcutaneously twice daily. Two days later, stimulation is initiated by intramuscular (IM) injections of HMG (Merional, IBSA, Germany) in a dose of 300 IU/day.

Follicular monitoring began from the ninth day of the cycle by serial vaginal ultrasonography and measurement of serum E2 levels. IM injections of 10000 IU HCG (Choriomon; IBSA, Germany) were injected when at least 2 follicles 18 mm were observed on ultrasonography.

Oocytes were retrieved 36 hours after hCG injection using a 17-gauge aspiration needle under transvaginal ultrasound guidance. The pelvis is evaluated with ultrasound to ensure that there is no internal bleeding.

After fertilization was confirmed when two polar bodies and two pronuclear were observed 18-20 hours after insemination, one to three grade A embryos were transferred at day 3 fertilization.

The luteal phase support was initiated from the day of oocyte retrieval for all patients with (Cyclogest 400 mg, Actavis pharmaceutical, UK) vaginal suppositories per day till the day of serum pregnancy test was done.

Serum β-hCG was performed 14 days after the embryo transfer to confirm chemical pregnancy. Clinical pregnancy was confirmed when there was an evidence of gestational sac, embryo and fetal heart activity at time of transvaginal ultrasound evaluation by the 6th week.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a history of one or more failed IVF cycles with three or less retrieved oocytes
2. No age limitation
3. Patients with an inadequate ovarian response in previous cycle
4. Low estradiol (E2) levels in response to ovarian stimulation in previous cycle
5. Lower number of retrieved oocytes in previous trials.

Exclusion Criteria:

1. Severe male factor (azospermia)
2. Hydrosalpinx
3. History of endometriosis
4. Endocrine or metabolic disorders
5. Follicle stimulating hormone (FSH) level > 15 mIU.
6. Antimullerian hormone (AMH)< 0.5 ng/ml
7. Any uterine causes of infertility e.g. septate uterus

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy | 4 weeks after embryo transfer
  Intrauterine gestational sac detection by transvaginal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt